CLINICAL TRIAL: NCT03310333
Title: Comparison Between Two Strategies of Induction in Case of Unfavourable Cervix After 12 Hours of Premature Rupture of Membranes (PROM) at Term: Cook Cervical Ripening + Oxytocine From 6 Hours Versus Dinoprostone Vaginal Insert
Brief Title: Cook Balloon Versus Propess After 12 Hours of Rupture of Membranes
Acronym: RUBAPRO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-352; 2017-A00811-52 (Other: 2017-A00811-52)
Record Dates: First submitted 2017-09-27; First posted 2017-10-16 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: PROM (Premature Rupture Of Foetal Membrane)
Keywords: PROM; Dinoprostone; cervical ripening device; oxytocin
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Dinoprostone

STUDY DESIGN:
Masking Description: open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cook cervical ripening (Experimental): the device is introduced by a resident or a doctor. No traction on the probe was done. It is left in place for maximum 12 hours. Oxytocin is added at the end of the first 6 hours even if device is fallen. An epidural analgesia can be started before or after the installation of oxytocin
  Interventions: Device: cook cervical pipening balloon
- Dinoprostone vaginal group (Active Comparator): the device is placed in vaginal fornix by the midwife for maximum 24 hours. If Propess ® is fallen before the first 12 hours, another one could be introduce if the cervix stayed unfavourable.
  After 24 hours, it is removed. If they are any contraction, oxytocin is started with or without epidural analgesic.
  Interventions: Drug: Propess® (dinoprostone)

INTERVENTIONS:
Drug: Propess® (dinoprostone) — The inclusion begins after 12 hours of PROM for a pregnant woman who has an unfavourable cervix and no B streptococcus. The case is discussed during the obstetric staff every morning.
  If the cervix is unfavourable (cervical Bishop's score <6), the information of the study is given to the patient and the consent collected.
  An antibiotic is started at the beginning of the inclusion by amoxicillin (or clindamycin in case of allergy of amoxicillin) to prevent choroamnionitis.
  Arms: Dinoprostone vaginal group
Device: cook cervical pipening balloon — • In dinoprostone vaginal group: the device is placed in vaginal fornix by the midwife for maximum 24 hours. If Propess ® is fallen before the first 12 hours, another one could be introduce if the cervix stayed unfavourable.
  Arms: Cook cervical ripening

SUMMARY:
The objective is to demonstrate the superiority of the strategy of labor induction by Cook® cervical ripening balloon between recommended strategy by dinoprostone (propess®) on the reduction of the time between cervical ripening and delivery in case of unfavorable cervix after 12 hours of PROM in term pregnant women.

DETAILED DESCRIPTION:
The inclusion begins after 12 hours of PROM for a pregnant woman who has an unfavourable cervix and no B streptococcus. The case is discussed during the obstetric staff every morning.

If the cervix is unfavourable (cervical Bishop's score <6), the information of the study is given to the patient and the consent collected.

An antibiotic is started at the beginning of the inclusion by amoxicillin (or clindamycin in case of allergy of amoxicillin) to prevent choroamnionitis.

After randomization, the patient is included in one of the two groups: Cook ® balloon or Propess ®.

* In the Cook cervical ripening balloon group: the device is introduced by a resident or a doctor. No traction on the probe was done. It is left in place for maximum 12 hours. Oxytocin is added at the end of the first 6 hours even if device is fallen. An epidural analgesia can be started before or after the installation of oxytocin
* In dinoprostone vaginal group: the device is placed in vaginal fornix by the midwife for maximum 24 hours. If Propess ® is fallen before the first 12 hours, another one could be introduce if the cervix stayed unfavourable.

After 24 hours, it is removed. If they are any contraction, oxytocin is started with or without epidural analgesic.

* The fetal heart rate is monitoring 30 minutes before and after the insertion of the device. After, the patient has a monitoring each 6 hours.
* Since the oxytocin is started, the monitoring is registered in continue until the delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women

  * 18 years old With a singleton live cephalic pregnancy ≥ 37+0 weeks Gestational age estimated from the first trimester ultrasound (realized between 11 and 13+6 weeks of gestation) PROM without spontaneous labour in the 12 hours after the rupture. The diagnostic of PROM is clinic or biologic (ActimProm® test).

Unfavourable cervix (Bishop's score < 6) Agreement of the patient after clear, loyal and appropriate information Subject covered by or having the rights to the French Social Security system

Exclusion Criteria:

* Vaginal infection by B streptococcus or in urinary sample during actual or anterior pregnancy Meconium fluid amniotic Contraindication of vaginal delivery (placenta praevia, …) Temperature > 38,2°C Suspicion of chorio-amnionitis among Newton requirements Intra-uterine growth restriction < 3rd percentile with Doppler abnormalities History of cesarean and uterine scare Suspected genital herpes infection Known VIH seropositivity (confirmed by blood serology) Fetus with suspected severe congenital abnormalities Pathological fetal heart rate (see appendix 1) Contra-indications to Propess®, Cook® Cervical Ripening Balloon, Oxytocin Women under guardianship or trusteeship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Time between the beginning of the induction of labor and the delivery | at day 1

SECONDARY OUTCOMES:
Time limits between the PROM and the beginning of induction | at day 1
Rate of delivery in the first 24 hours | at day 1
Application time of Cook® balloon | at day 1
Application time of Propess® | at day 1
Time between labour induction and vaginal delivery | at day 1
Rate of vaginal delivery with and without extraction | at day 1
Rate of cesarean | at day 1
Rate of delivery hemorrhage | at day 1
Bischop score when Cook balloon is fallen or retry | at day 1
Rate of balloon present after 12 hours | at day 1
Rate of anomaly of fetal heart rate leading stop of dinoprostone | at day 1
Rate of epidural analgesia | at day 1
Time to obtain active labour | at day 1
Time to obtain complete cervix dilatation | at day 1
Rate of fever during the labour | at day 1
Rate of uterine hyperkinesias | at day 1
Rate of clinic chorio-amnionitis defined by Newton criteria | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Denis GALLOT, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Devillard E, Delabaere A, Rouzaire M, Pereira B, Accoceberry M, Houlle C, Dejou-Bouillet L, Bouchet P, Gallot D. Induction of labour in case of premature rupture of membranes at term with an unfavourable cervix: protocol for a randomised controlled trial comparing double balloon catheter (+oxytocin) and vaginal prostaglandin (RUBAPRO) treatments. BMJ Open. 2019 Jun 20;9(6):e026090. doi: 10.1136/bmjopen-2018-026090. PMID 31227530